CLINICAL TRIAL: NCT01446354
Title: Does the Intraoperative Thromboelastometry-guided Coagulation Management Reduce the Administration of Allogeneic Blood Products in Cardiac Surgery With the Help of Hypothermic Cardiac Arrest? A Retrospective Data Analysis
Brief Title: Goal-orientated Coagulation Management in Hypothermic Cardiac Arrest Surgery
Status: Completed | Type: Observational
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Principal Investigator, Daniel Bolliger, Principal Investigator, University Hospital, Basel, Switzerland
Other Study IDs: 347/10
Record Dates: First submitted 2011-09-29; First posted 2011-10-05 (Estimated); Last update posted 2012-10-24 (Estimated); Status verified 2012-10

CONDITIONS: Cardiac Arrest
Keywords: Blood component transfusion; Hypothermic
MeSH Terms: conditions — Heart Arrest; Hypothermia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Cardiac surgery with HCA: Patients undergoing cardiac surgery with the help of hypothermic cardiac arrest for pathologies of the proximal aorta

SUMMARY:
Cardiac surgery including hypothermic cardiac arrest (HCA) commonly involves perioperative transfusion of allogeneic blood products which is associated with increased morbidity and mortality. In this retrospective analysis, the investigator aimed to evaluate the effect of a thromboelastometry-guided treatment algorithm promoting fibrinogen concentrate as first line hemostatic agent on the perioperative use of allogeneic blood products.

DETAILED DESCRIPTION:
The investigators will analyze the data of patients undergoing elective and emergent surgical procedures involving the ascendent aorta and/or the aortic arch with the help of HCA from January 2009 to June 2011.

The investigators will collect and document baseline characteristics, the use of thromboelastometry, thromboelastometric data, and perioperative laboratory data. In addition, the investigators will evaluate perioperative bleeding from mediastinal drainages, perioperative use of blood and hemostatic products, and the adverse events within the hospitalisation including re-exploration, renal impairment, myocardial infarction, severe brain injury, and death.

ELIGIBILITY:
Inclusion Criteria:

* Cardiac surgery with HCA due to pathology of the proximal aorta from January 2009 until June 2011

Exclusion Criteria:

* none

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients undergoing cardiac surgery with the help of hypothermic cardiac arrest
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2011-01; Primary Completion 2011-12 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
Transfusion of allogeneic blood products | within 24 hours including surgery

SECONDARY OUTCOMES:
Proportion of patients without allogeneic blood products | 24 hours including surgery
Adverse events | within 24 hours including surgery
  Adverse events include: renal impairment (RIFLE criteria), stroke, severe neurologic impairment, myocardial infarction, death, re-exploration

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Bolliger, PD Dr., Principal Investigator — University Hospital, Basel, Switzerland
Locations (1):
- University Hospital Basel, Department of Anesthesia and Intensive Care Medicine, Basel, Canton of Basel-City, Switzerland